CLINICAL TRIAL: NCT01815957
Title: Impact of Ranalozine on Coronary Microcirculatory Resistance- A Prospective Single Center Study to Evaluate the Effect of Ranalozine in Microcirculatory Resistance (MICRO Study)
Brief Title: Impact of Ranolazine on Coronary Microcirculatory Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-069 MICRO Study
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Coronary Microcirculation; Coronary Artery Disease; Myocardial Disease; Ischemia
Keywords: coronary microcirculation; coronary artery disease; myocardial disease; ischemia
MeSH Terms: conditions — Coronary Artery Disease; Cardiomyopathies; Ischemia | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranalozine (Experimental): After enrollment in the study, participants will initiate Ranolazine for 4 weeks. The participant's usual anti-anginal medication regimen will be continued unchanged throughout study duration. Patients will receive Ranolazine 500 mg orally twice daily for 1 week, and the dose will be increased to 1,000 mg twice daily for an additional 3 weeks if tolerated.
  Interventions: Drug: Rnalozine

INTERVENTIONS:
Drug: Rnalozine — . After enrollment in the study, participants will initiate Ranolazine for 4 weeks. The participant's usual anti-anginal medication regimen will be continued unchanged throughout study duration. Patients will receive Ranolazine 500 mg orally twice daily for 1 week, and the dose will be increased to 1,000 mg twice daily for an additional 3 weeks if tolerated.
  Other Names: Ranexa; Ranalozine

SUMMARY:
This study is being done to determine if Ranolazine treatment improves coronary microcirculation function among patients with coronary microcirculation dysfunction. We are also looking to learn if symptomatic improvement of chest pain during treatment with Ranalozine is related to improved coronary microcirculation function.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with subjective symptoms of ischemia without flow limiting angiographic CAD (<50% epicardial coronary stenosis) and abnormal IMR (>20 U).
* Definition of ischemia (any one):

  * chest pain with dynamic ischemic ECG changes (t wave inversions or > 1 mm ST depressions
  * Exercise treadmill testing induced chest pain with ≥1 mm of downsloping or flat ST segment depression during exercise or recovery; ≥2 mm of ischemic ST depression at a low workload (stage 2 or less or ≤130 beats/min); early onset (stage 1) or prolonged duration (>5 min) of ST depression; multiple leads (>5) with ST depression
  * Nuclear stress perfusion defect > 10%
  * Stress echocardiogram with stress induced wall motion abnormality

Exclusion Criteria:

* - Age < 18 yrs
* Flow Limiting epicardial CAD >50%
* Life expectancy < 6 months
* Recent (<1 week) myocardial infarction or positive biomarkers
* Severe aortic stenosis
* Contraindications to IMR testing including inability to utilize antithrombotic therapy and/or intravenous adenosine
* Contraindications to Ranolazine therapy:
* Patients with known hepatic insufficiency, prolonged QT or renal failure (GFR < 60)
* use of drugs that inhibit CYP3A such as diltiazem, verapamil, ketoconazole, macrolides and HIV protease inhibitors
* Pregnancy, breastfeeding
* Patients taking drugs which prolong QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bina Ahmed, MD, Principal Investigator — Assistant Professor, IM Div Cardiology
Locations (1):
- University of New Mexico Health Science Center, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Publication:
  Title: Impact of ranolazine on coronary microvascular dysfunction (MICRO) study Published in Cardiovascular Revascularization Medicine: Volume 18, Issue 6, September 2017, Pages 431-435
  Please refer to Table 1 for the Baseline Demographic Variables
Period: Overall Study
Arm/Group | Ranalozine
Started | 7
Completed | 0
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Ranalozine
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 57.6 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Relative Change in the Index of Microcirculatory Resistance Before and After Ranolazine Therapy
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ranalozine
Number analyzed (Participants) | 7
Participants | 7

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Ranalozine: Ranolazine 500 mg BID
- Ranalozine Titration: After 7 days, 1000 mg BID
Arm/Group | Ranalozine | Ranalozine Titration
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT01815957/Prot_000.pdf
  • Informed Consent Form (2015-03-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT01815957/ICF_001.pdf